CLINICAL TRIAL: NCT02983890
Title: Dicloxacillin: Clinical Relevance of Drug-drug Interactions by Induction of Drug Metabolizing Enzymes.
Brief Title: Dicloxacillin: Clinical Relevance of Drug-drug Interactions by Induction of Drug Metabolism.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Per Damkier (Other)
Responsible Party: Sponsor-Investigator, Per Damkier, Professor, head consultant, MD, ph.d., Odense University Hospital
Organization: Odense University Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AKF-388
Record Dates: First submitted 2016-11-30; First posted 2016-12-06 (Estimated); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Healthy
MeSH Terms: interventions — Dicloxacillin; Anti-Bacterial Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm of study1 (Active Comparator): Dicloxacillin tablets.
  Interventions: Drug: Dicloxacillin
- Arm of study 2 (Placebo Comparator): No treatment
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Dicloxacillin — Tablets containing dicloxacillin are taken 500mg 2x 3 times per day, for 10 days. Followed by test-day nr 1 at day 11.
  Both arms receives both treatments, randomly assigned
  Other Names: antibiotics
  Arms: Arm of study1
Drug: Placebos — No drug are taken for 10 days. Non-blinded. Followed by test-day nr 1 at day 11.
  Both arms receives both treatments, randomly assigned
  Arms: Arm of study 2

SUMMARY:
This trial is conducted as a cocktail-study namely an open-label, randomized, two-sequence, two-period crossover, cocktail study where a combination of cocktail-drugs is used to illustrate whether or not, or to what degree dicloxacillin affects the level of activity of the 5 most important CYP enzymes and therefore plays a potentially decisive role in serious drug-drug interactions.

DETAILED DESCRIPTION:
Given knowledge explains dicloxacillin and the drug warfarin to be a potential dangerous drug drug interaction because the effects of warfarin is downregulated to a degree as to where it might cause patients to have thrombotic events.

A potential explanation to this is namely dicloxacillin increases the activity of certain drug metabolising enzymes metabolising warfaring which in turn decreases the concentration of the drug in the blood and the therapeutic effect.

Cocktail study is the golden standard to investigate as to whether there is changes is P450 enzymes as a result of drug-drug interactions.

The cocktail consists of Midazolam, omeprazole, tolbutamide, caffein and dextromethorphan which is well known markers for these enzymes. These markers are safe, have specific (enzyme) metabolism and has been used in several studies with no Serious Adverse reactions reported.

By measuring the Concentration of the drug and its metabolites in plasma / Urine before and after treatment with dicloxacillin we will estimate AUC (area under the curve) and test our hypothesis/primary end point of whether there is change in AUC for Tolbutamide (CYP2C9)

ELIGIBILITY:
Inclusion Criteria:

* Are you in a general healthy condition?; questions asked; Are you healthy in general? 2; Do you have any chronic diseases? 3; Are you taking any medications regularly? 4, Are you taking any medications periodically . 5; Are you taking nutrition supplements, "nature-medicine" or over-the-counter drugs
* BMI; range; 18,5-29,9 kg/m2
* eGFR(estimated glomerular filtration rate), ALAT(alanine aminotransferase), bilirubin, hæmoglobin og HbA1c, should be within normal limits or without clinically significantly deviation from these.
* Non-Smoker

Exclusion Criteria:

* Hypersensitivity to applied medications. Known allergy to penicillin or type 1-reaction to cefalosporins.
* Known allergy to sulfonamides
* Clinically relevant intake of receipt-required medication, over-the-counter medication or nutritional supplements.
* Chronic or daily intake of alcohol.
* Participation in other Intervention-studies

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2016-10-06 (Actual); Primary Completion 2017-04-05 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
AUC(area under the curve) for tolbutamid (CYP2C9), as a result of dicloxacillin-treatment | Pharmacological outcome measures at t=0 predose and postdose; 0.5,1,2,3,4,6,8,10,12,24.
  AUC measurements giving an estimate of activity og the relevant enzymes.

SECONDARY OUTCOMES:
*AUC(area under the curve) for midazolam (CYP3A4) and dextromethorphan (CYP1A2) omeprazole (CYP2C19) and caffein (CYP1A2) | Pharmacological outcome measures at t=0 predose and postdose; 0.5,1,2,3,4,6,8,10,12,24.
T(max) | Pharmacological outcome measures at t=0 predose and postdose; 0.5,1,2,3,4,6,8,10,12,24.
  The amount of time that the drug is present at the maximum concentration in serum.
C(max) (peak plasma concentration) | Pharmacological outcome measures at t=0 predose and postdose; 0.5,1,2,3,4,6,8,10,12,24.
  The peak serum concentration of a therapeutic drug.
Clearance | Pharmacological outcome measures at t=0 predose and postdose; 0.5,1,2,3,4,6,8,10,12,24.
  The volume of plasma from which the drug is completely removed per unit time. Reflects rate of drug elimination divided by plasma concentration.

CONTACTS AND LOCATIONS:
Overall Officials: Per Damkier, Ph.d., Principal Investigator — Assosiated to department of biochemistry and pharmacology at University of southern denmark, Odense
Locations (1):
- Klinisk Biokemisk Farmakologi syddansk universitet, Odense, Funen, Denmark

IPD SHARING:
Plan to Share IPD: No